CLINICAL TRIAL: NCT04742569
Title: Wearable Diagnostic for Detection of COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: ClinOne, Inc. (Industry)
Collaborators: BioIntelliSense, Inc (Unknown); Phillips North America, LLC (Unknown); University of Colorado, Denver (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 1294415
Record Dates: First submitted 2021-01-14; First posted 2021-02-08 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: Recent known exposure to COVID-19; Asymptomatic; Early COVID-19 Symptoms
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1- Exposed/Early Symptomatic: The population identified for this study includes subjects who request COVID-19 testing in response to a concern for recent COVID-19 exposure and/or concern of COVID-19-like related symptoms. We will recruit and enroll patients through public facing websites, clinic and pharmacy vaccination schedules and on-site vaccination marketing.
  For the population with recent COVID-19 exposure and/or concern of COVID-19-like related symptoms, population identification includes subjects who visit eTrueNorth's https://www.doineedacovid19test.com/ website where subjects have access to over 7,500 testing site locations across the nation. Otherwise, individuals seeking COVID-19 testing will be directed to the ClinOne, Inc. website for information regarding the Wearable Diagnostic for Detection of COVID-19 Infection study contact information for study participation, enrollment into the study using eConsent, and will receive a BioSticker wearable kit by express mail the next day.
- CoHort 2- Pfizer or Moderna Vaccine: Secondly, the other population identified for this study includes subjects who are scheduled for the first and second dose of the mRNA-based Pfizer/BioNTech and Moderna vaccine series. For the population seeking the mRNA-based Pfizer/BioNTech and Moderna vaccine series, we will recruit and enroll patients through public-facing websites, clinic, and pharmacy vaccination schedules, and on-site vaccination marketing

SUMMARY:
The goals of this study are 1) to validate the use of a wearable diagnostic capability and software as a medical device (SaMD) algorithm for the pre or early-symptomatic detection of COVID-19 infection, 2) assess the wearable device on the subjects, and 3) ensure data are collected, securely stored, and easily read and interpreted by non-laboratory personnel.

DETAILED DESCRIPTION:
This is an open label iterative study designed to calibrate the algorithm to maximize its test characteristics. The sample size is derived from the minimum number of COVID-19 subjects required to evaluate algorithm sensitivity and specificity. A sample size of 200 true positive COVID-19 infections is anticipated to assess device predictive analytics. Assuming a six-month enrollment period, a 15 percent patient lost to follow-up rate, and a positive COVID-19 infection rate of 10 percent within the study population, a sample size of 2,352 subjects will be enrolled in this prospective study.

Primary Outcomes: The primary outcomes of interest are performance of the BioSticker multiparameter vital signs wearable and the sensitivity of the BioCloud-based algorithms in detecting early onset of active COVID-19 related signs and symptom in subjects prior to or coincident with a positive COVID-19 diagnostic test and the specificity of the BioSticker algorithms in distinguishing positive diagnosis of infection from negative diagnosis of infection among subjects. COVID-19 infection will be confirmed by both participant affirmation and diagnostic laboratory testing. Additional primary outcome is the intuitive presentation of affirmative diagnostic results from the BioSticker early detection algorithm(s).

Secondary Outcomes: The secondary outcomes of interest include correlation of biometric data indicators to individual-level experiential feedback reported through participant symptom-tracking and diagnostic questionnaires.

ELIGIBILITY:
Cohort 1- Exposed/ Early Symptomatic Group

Inclusion Criteria:

1. age 18 or older;
2. able to follow the study device wear instructions per the Instructions for Use;
3. no positive viral test within 60 days prior to enrollment; and
4. willing and able to provide written, informed consent.

Exclusion Criteria:

1. pregnant or breastfeeding;
2. wearing a defibrillator or pacemaker;
3. known or suspected cardiac dysrhythmias
4. known or suspected allergy to adhesives;
5. chronic daily use of non-steroidal anti-inflammatory medications (NSAIDs) and antipyretic medications
6. open wounds or infected, irritated, scarred, or inflamed areas of skin on the upper chest preventing placement of the biosensor; and
7. current or planned use of either an investigation pharmaceutical or an investigational device during the study.

Cohort 1- Vaccine Group

Inclusion Criteria:

Subjects seeking the mRNA-based Pfizer/BioNTech and Moderna vaccine series are eligible for the study if they are:

1. Age 18 or older; 12 years of age -17 years of age are approved to participate in the vaccine Cohort portion of the study.
2. scheduled to receive their first and second dose of the Pfizer/BioNTech or Moderna COVID-19 vaccine
3. able to follow the study device wear instructions per the Instructions for Use;
4. no positive viral test within 60 days prior to enrollment; and
5. willing and able to provide written, informed consent.
6. Willing and able to take an oral temperature

Exclusion Criteria:

Potential subjects seeking the mRNA-based Pfizer/BioNTech and Moderna vaccine series will be excluded from the study if they are or have any of the following:

1. pregnant or breastfeeding;
2. wearing a defibrillator or pacemaker;
3. known or suspected cardiac dysrhythmias
4. known or suspected allergy to adhesives;
5. chronic daily use of non-steroidal anti-inflammatory medications (NSAIDs) and antipyretic medications
6. open wounds or infected, irritated, scarred, or inflamed areas of skin on the upper chest preventing placement of the biosensor; and
7. current or planned use of either an investigation pharmaceutical or an investigational device during the study.
8. previously fully vaccinated subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort 1- Exposed/Early Symptomatic Group All adult subjects seeking a COVID-19 test and meeting enrollment criteria will be offered enrollment into this study.
  The Inclusion Criteria are:
  1. Adults - 18 years of age and older
  2. Both genders, all races and ethnic groups
  3. English speaking adult subjects only
  Cohort 2- Vaccine Group:
  Potential subjects seeking the mRNA-based Pfizer/BioNTech and Moderna vaccine
  1. Subjects who are scheduled to receive the COVID vaccination series through local and national clinics, health systems and pharmacies.
  2. Subjects who become aware of the study through public notices, postings, and advertisements, and other marketing efforts.
Sampling Method: Probability Sample
Enrollment: 790 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
The primary outcome of interest are performance of the BioSticker, a medical grade multi-parameter wearable biosensor. | 14 days
  Biometric data will be measured for 14 days using the application of the BioSticker on the upper left side of the chest.
The primary outcome of interest are performance of the BioSticker, a medical grade multi-parameter wearable biosensor. | 14 days
  Vital Signs measurements will be collected for 14 days using the application of the BioSticker on the upper left side of the chest.
The primary outcome of interest are performance of the BioSticker wearable for detecting early onset of active COVID-19 related symptoms. | 14 days
  Symptom tracking data will be collected through daily questionnaires for 14 consecutive days, administered through ClinOne. Health data known to be associated with COVID-19 risk and severity, including comorbid conditions, risk factors, and demographic data will be collected from subjects during screening and enrollment via the ClinOne study website.
The primary outcome of interest is the sensitivity of the BioCloud-based algorithms in detecting early onset of active COVID-19. | 14 days
  BioSticker sensor data will be time-stamped and annotated against clinical events (e.g., fever, cough), symptom progression data, and other indicators of infection as they are identified. Weighting coefficients for predictive algorithms will be tuned and algorithms will be iteratively refined using machine learning methods and small batches of data anticipated to include between 20 and 50 positive cases per set, and validated against sensor data obtained from COVID-19-negative subjects.

SECONDARY OUTCOMES:
The secondary outcomes of interest include correlation of biometric data indicators to patient reported symptoms. | 14 days
  Individual-level experiential feedback will be reported through participant symptom- tracking and diagnostic questionnaires for 14 consecutive days.

CONTACTS AND LOCATIONS:
Overall Officials: James Mault, MD, Principal Investigator — BioIntelliSense, Inc
Locations (1):
- ClinOne, Inc, Greenwood Village, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buitrago-Garcia D, Egli-Gany D, Counotte MJ, Hossmann S, Imeri H, Ipekci AM, Salanti G, Low N. Occurrence and transmission potential of asymptomatic and presymptomatic SARS-CoV-2 infections: A living systematic review and meta-analysis. PLoS Med. 2020 Sep 22;17(9):e1003346. doi: 10.1371/journal.pmed.1003346. eCollection 2020 Sep. PMID 32960881
- [Result] Kucirka LM, Lauer SA, Laeyendecker O, Boon D, Lessler J. Variation in False-Negative Rate of Reverse Transcriptase Polymerase Chain Reaction-Based SARS-CoV-2 Tests by Time Since Exposure. Ann Intern Med. 2020 Aug 18;173(4):262-267. doi: 10.7326/M20-1495. Epub 2020 May 13. PMID 32422057
- [Result] Natarajan A, Su HW, Heneghan C. Assessment of physiological signs associated with COVID-19 measured using wearable devices. NPJ Digit Med. 2020 Nov 30;3(1):156. doi: 10.1038/s41746-020-00363-7. PMID 33299095
- [Result] Ra SH, Lim JS, Kim G, et al. Thorax Epub ahead of print: 2020 September 22; doi:10.1136/ thoraxjnl-2020-215042
- [Result] Rudolph JL, Halladay CW, Barber M, McConeghy KW, Mor V, Nanda A, Gravenstein S. Temperature in Nursing Home Residents Systematically Tested for SARS-CoV-2. J Am Med Dir Assoc. 2020 Jul;21(7):895-899.e1. doi: 10.1016/j.jamda.2020.06.009. Epub 2020 Jun 9. PMID 32674815